CLINICAL TRIAL: NCT07114536
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate theEffects of Calcium Alpha-Ketoglutarate Supplementation on BiologicalAging, Physical Performance, and Metabolic Health in Middle-Aged andOlder Adults
Brief Title: Evaluation of the Efficacy of Calcium a -Ketoglutarate(AKG-Ca) in Improving Human Aging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Hygieia Biotech Co., Ltd (Industry)
Collaborators: Zhejiang Chinese Medical University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Evaluation of AKG-Ca on Aging
Record Dates: First submitted 2025-07-31; First posted 2025-08-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-08

CONDITIONS: Aging
Keywords: a-ketoglutaric acid; Phenoage*age; Healthy aging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: calcium-a-ketoglutarate (Experimental): The experimental group subjects took four Ca-AKG tablets (0.5 g/tablet) daily.
  Interventions: Dietary Supplement: Calcium-a-ketoglutarate
- Control group: starch (Placebo Comparator): Placebo-controlled group subjects took four starch placebo tablets (0.5g/tablet) daily.
  Interventions: Other: Placebo(starch)

INTERVENTIONS:
Dietary Supplement: Calcium-a-ketoglutarate — Description: Participants in the intervention group will receive oral calcium alpha-ketoglutarate (CaAKG) in granular tablet form. Each tablet contains 0.5 grams of CaAKG.Participants will take two tablets twice daily (morning and evening). The total daily dose is 2 grams. The intervention period will last for 12 weeks. CaAKG is a stabilized form of alpha-ketoglutarate that enhances bioavailability and provides supplemental calcium. The tablets are identical in appearance and texture to those in the placebo group to maintain blinding.
  Arms: Intervention group: calcium-a-ketoglutarate
Other: Placebo(starch) — Participants in the placebo group will receive oral tablets identical inappearance and texture to the CaAKG tablets, but containing starch with no active calciumalpha-ketoglutarate. Each tablet weighs 0.5 grams. Participants will take two tablets twicedaily (morning and evening), for a total daily intake of 2 grams. The placebo tablets arepackaged and administered in the same manner as the CaAKG tablets to ensure blindingthroughout the 12-weekintervention period.
  Arms: Control group: starch

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial aims to evaluate the effects of calcium alpha-ketoglutarate (CaAKG) supplementation on biological aging and age-related health indicators in middle-aged and older adults. Alpha-ketoglutarate (AKG), a key intermediate in the Krebs cycle, has been investigated for its potential role in modulating aging-related metabolic and cellular pathways. Due to the poor oral bioavailability of free AKG, its stabilized form-calcium alpha-ketoglutarate (CaAKG)-is used to enhance absorption and additionally provides calcium supplementation benefits. At the population level, there is currently a lack of systematic assessment studies on the effects of CaAKG on human ageing-related indicators.

The study will recruit generally healthy adults aged 45 to 75 years. Participants will be randomly assigned to receive either CaAKG or a placebo daily for 12 weeks. The primary objective is to assess changes in biological aging, as measured by PhenoAge. Secondary outcomes include changes in physical performance, inflammatory markers, glucose and lipid metabolism, ageing-related gene expression, and self-reported quality of life.

This trial is designed to provide evidence on the efficacy and safety of CaAKG as a potential dietary intervention to support healthy aging. All participants will undergo pre- and post-intervention assessments. The study has been reviewed and approved by Medical Ethics Committee of Zhejiang Chinese Medical University, and informed consent will be obtained from all participants prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40-75 years old, no gender restrictions.
2. Has not taken any other anti-ageing research products in the past two months.
3. Able to use a smartphone.
4. Informed consent, voluntarily signed informed consent form, and agreed to participate in all visits and treatments in accordance with the trial protocol.

Exclusion Criteria:

1. Patients with cardiovascular disease, severe/uncontrolled hypertension, rheumatic heart disease, congenital heart disease, deep vein thrombosis, or pulmonary embolism .
2. Patients with Type I/Type II diabetes (treated with oral metformin or insulin) or diabetes complications .
3. Patients with cancer or who have undergone surgery, systemic drug therapy, or radiation therapy within the past 3 years.
4. Chronic obstructive pulmonary disease (COPD), severe asthma (requiring daily medication).
5. Multiple sclerosis, autoimmune/immunodeficiency disorders.
6. Recent history of sepsis or infection (hospitalisation within the past 3 months).
7. Any mental illness or neurodegenerative disease.
8. Any metallic implants in the body.
9. Hepatitis/cirrhosis.
10. Severe kidney disease (GFR <30 mL/min/1.73 m²).
11. Suffering from other conditions deemed unsuitable for participation in this trial (as determined by the investigator).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in PhenoAge from Baseline to Week 12 | Baseline and Week 12
  Phenotypic Age (PhenoAge) is a composite biomarker-based estimate of biological age. The primary outcome is the change in PhenoAge from baseline to the end of the 12-week intervention period. PhenoAge will be calculated using the algorithm developed by Levine et al. (2018), based on a validated mortality risk model.

SECONDARY OUTCOMES:
Change in Calcium Content of Bone | Baseline and Week 12
  The calcium content of bone will be measured at baseline and at Week 12 to evaluate changes resulting from CaAKG supplementation. Bone calcium will be assessed using dual-energy X-ray absorptiometry (DXA) with mineral content analysis at specific skeletal sites. The primary metric is the change in bone calcium content (mg/cm2 or mg) over the 12-week intervention period.
Change in β-Galactosidase Activity | Baseline and Week 12
  β-Galactosidase activity will be measured in serum collected at baseline and at Week 12.
Change in Age-related Gene Expression | Baseline and Week 12
  e.g., SIRT1~7、TERT/TERC、p21(CDKN1A)、p16INK4a(CDKN2A)、PDGFRB、PLOD1、MAP4K4、NFKBIA、GFAP、F2RL3、HERPUD1、PPPIR15A、PCBP1、TFAM、MMP7
Change in Grip strength | Baseline,12-week study
  The change in Grip strength (kg) of 30 volunteers before and after the intervention was measured.
Change in body Weight | Baseline and Week 12
  The change in body weight (kg) of 30 volunteers before and after the intervention was measured.
Change in body mass index(BMl) | Baseline and Week 12
  The change in Body Mass Index (BMl) kg/m2 of 30 volunteers before and after the intervention was measured.
Change in body fat mass | Baseline and Week 12
  The change in body fat mass(kg) of 30 volunteers before and after the intervention was measured.
Change in alkaline phosphatase (ALP) | Baseline and Week 12
  The change in alkaline phosphatase (ALP) in U/L of 30 volunteers before and after the intervention was measured.
Change in body fat percentage | Baseline and Week 12
  The change in body fat percentage (%) of 30 volunteers before and after the intervention was measured.
Change in fat-free mass | Baseline and Week 12
  The change in fat-free mass(kg) of 30 volunteers before and after the intervention was measured.
Change in muscle mass | Baseline and Week 12
  The change in muscle mass (kg) of 30 volunteers before and after the intervention was measured.
Change in body water | Baseline and Week 12
  The change in body water (kg) of 30 volunteers before and after the intervention was measured.
Change in blood creatinine (CREA) | Baseline and 12-week study.
  The change in blood creatinine (CREA) in mol/L of 30 volunteers before and after the intervention was measured.
Change in protein | Baseline and Week 12
  The change in protein (kg) of 30 volunteers before and after the intervention was measured.
Change in inorganic salts | Baseline and Week 12
  The change in inorganic salts (kg) of 30 volunteers before and after the intervention was measured.
Change in TotalT lymphocytes (CD3+) | Baseline and Week 12
  The change in TotalT lymphocytes (CD3+) (cells/μl) of 30 volunteers before and after the intervention was measured.
Change in helper T cells(cD4+) | Baseline and Week 12
  The change in helper T cells (CD4+) (cells/μl) of 30 volunteers before and after the intervention was measured.
Change in cytotoxicT cells(CD8+) | Baseline and Week 12
  The change in cytotoxic T cells (CD8+)(cells/μL) of 30 volunteers before and after the intervention was measured.
Change in Glycated haemoglobin (HbAlc) | Baseline and Week 12
  The change in Glycated haemoglobin (HbA1c) (%) of 30 volunteers before and after the intervention was measured.
Change in Fasting blood glucose | Baseline and Week 12
  The change in Fasting blood glucose (mmol/L) of 30 volunteers before and after the intervention was measured.
Change in Fasting insulin | Baseline and Week 12
  The change in Fasting insulin (pmol/L) of 30 volunteers before and after the intervention was measured.
Change in Physical activity questionnaire Scores | Baseline and Week 12
  International Physical Activity Questionnaire - Long Form (IPAQ-LF). At baseline and 12 weeks, measure changes in participants' Physical activity questionnaire scores. There is no fixed upper or lower limit to the total score, but scores at different activity intensities (walking, moderate intensity, high intensity) can be accumulated based on metabolic equivalents (MET-min/week). Higher score: Reflects the greater the total amount of physical activity an individual has engaged in in the past week.
Change in number of finger taps in one minute | Baseline and Week 12
  The change in number of finger taps in one minute of 30 volunteers before and after the intervention was measured.

OTHER OUTCOMES:
Change in Gut Microbiota | Baseline, 12-week study
  16S rRNA sequencing
Change in Urea (UREA) | Baseline and 12-week study
  The change in Urea (UREA) in mmol/L of 30 volunteers before and after the intervention was measured.
Change in Blood routine test | Baseline, 12-week study
  Blood routine examination indicators
Change in Total Bilirubin | Baseline and 12-week study
  The change in Total Bilirubin(μmol/L) of 30 volunteers before and after the intervention was measured.
Changes in SF-36 Questionnaire Scores | Baseline, 12-week study
  36-Item Short Form Health Survey. At baseline and 12 weeks, measure changes in participants' SF-36 questionnaire scores. The score range for each dimension of the SF-36 questionnaire is 0~100 points, with 0 representing the worst health status in the dimension and 100 representing the best. The composite score (PCS and MCS) is a mean of 50, and the higher the score, the better the physical or mental health, such as strong physical function and emotional stability; Lower scores indicate more serious health problems, such as pain, functional limitations, or psychological distress.
Change in High-sensitivity C-reactive protein(hs-CRP) | Baseline and Week 12
  The change in High-sensitivity C-reactive protein(hs-CRP) in mg/L of 30 volunteers before and after the intervention was measured.
Change in Direct bilirubin | Baseline,12-week study
  The change in Direct bilirubin(μmol/L) of 30 volunteers before and after the intervention was measured.
Change in Indirect bilirubin | Baseline, 12-week study
  The change in Indirect bilirubinlumol/L) of 30 volunteers before and after the intervention was measured.
Change in Total bile acid | Baseline,12-week study
  The change in Total bile acid(μmol/L) of 30 volunteers before and after the intervention was measured.
Change in Albumin | Baseline, 12-week study
  The change in Albumin(g/L) of 30 volunteers before and after the intervention was measured.
Change in Globulin | Baseline,12-week study
  The change in Globulin(g/L) of 30 volunteers before and after the intervention was measured.
Change in tumour necrosis factor (TNF-a) | Baseline and 12-week study
  The change in tumour necrosis factor (TNF-a) in pg/mL of 30 volunteers before and after the intervention was measured.
Change in interleukin-2 (lL-2) | Baseline and 12-week study
  The change in interleukin-2 (lL-2) in pg/mL of 30 volunteers before and after the intervention was measured.
Change in Interleukin-6 | Baseline and 12-week study
  The change in Interleukin-6 (lL-6) in pg/mL of 30 volunteers before and after the intervention was measured.
Change in Interleukin-8 (lL-8) | Baseline and 12-week study
  The change in Interleukin-8 (lL-8) in pg/mL of 30 volunteers before and after the intervention was measured.
Change in interleukin-10 (lL-10) | Baseline and 12-week study
  The change in interleukin-10 (lL-10) in pg/mL of 30 volunteers before and after the intervention was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Li Jiaomei, Study Chair — Zhejiang Chinese Medical University
Locations (1):
- Zhejiang Chinese Medicine University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Protect volunteers' personal health data and personal privacy.

REFERENCES:
- [Result] Demidenko O, Barardo D, Budovskii V, Finnemore R, Palmer FR, Kennedy BK, Budovskaya YV. Rejuvant(R), a potential life-extending compound formulation with alpha-ketoglutarate and vitamins, conferred an average 8 year reduction in biological aging, after an average of 7 months of use, in the TruAge DNA methylation test. Aging (Albany NY). 2021 Nov 30;13(22):24485-24499. doi: 10.18632/aging.203736. Epub 2021 Nov 30. PMID 34847066
- [Result] Sandalova E, Goh J, Lim ZX, Lim ZM, Barardo D, Dorajoo R, Kennedy BK, Maier AB. Alpha-ketoglutarate supplementation and BiologicaL agE in middle-aged adults (ABLE)-intervention study protocol. Geroscience. 2023 Oct;45(5):2897-2907. doi: 10.1007/s11357-023-00813-6. Epub 2023 May 23. PMID 37217632
- [Result] Liu Z, Kuo PL, Horvath S, Crimmins E, Ferrucci L, Levine M. A new aging measure captures morbidity and mortality risk across diverse subpopulations from NHANES IV: A cohort study. PLoS Med. 2018 Dec 31;15(12):e1002718. doi: 10.1371/journal.pmed.1002718. eCollection 2018 Dec. PMID 30596641
- [Result] Liu C, Hua L, Xin Z. Synergistic impact of 25-hydroxyvitamin D concentrations and physical activity on delaying aging. Redox Biol. 2024 Jul;73:103188. doi: 10.1016/j.redox.2024.103188. Epub 2024 May 10. PMID 38740004

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT07114536/Prot_SAP_ICF_000.pdf